CLINICAL TRIAL: NCT01625819
Title: Exploring Tai Chi as a Behavioral Intervention for Heart Failure Patients
Brief Title: Exploring Behavioral Interventions to Improve Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura S. Redwine, PhD, Assistant Adjunct Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01HL096784-01A2 (NIH)
Record Dates: First submitted 2012-04-18; First posted 2012-06-21 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure
Keywords: Tai Chi
MeSH Terms: conditions — Heart Failure | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tai Chi (Experimental): 32 1-hour group sessions of Tai Chi instruction
  Interventions: Behavioral: Tai Chi
- Resistance Band (Active Comparator): 32 1-hour bi-weekly group sessions of Resistance Band exercises
  Interventions: Behavioral: Resistance Band
- Health Education (Placebo Comparator): 32 1-hour bi-weekly group sessions of health education
  Interventions: Behavioral: Health Education
- Care as Usual (No Intervention): Receive usual cardiology care for 4 months between pre- and post-treatment testing

INTERVENTIONS:
Behavioral: Tai Chi — 32 1-hour bi-weekly group sessions of Tai Chi instruction
  Arms: Tai Chi
Behavioral: Resistance Band — 32 1-hour bi-weekly group sessions of Resistance Band exercises
  Arms: Resistance Band
Behavioral: Health Education — 32 1-hour bi-weekly group sessions of health education
  Arms: Health Education

SUMMARY:
The objective of this research is to compare Tai Chi versus Resistance Exercise, Health Education and usual care for changes in cardiac functional capacity measured for ability of the heart to pump by measuring ejection fraction (EF), end systolic and diastolic volumes in heart failure (HF) patients. Also measured will be changes in physical function measured by walking speed and distance in the 6-min walk task, work performed during a bicycle task, and changes in daily physical activity. The investigators will compare groups for altered well-being including: depression, sleep disturbances, fatigue, mindfulness, spirituality and quality of life. In addition the investigators will compare groups for altered vascular and pro-inflammatory markers, catecholamines, and autonomic function at rest and in response to the bicycle task. Also, the investigators will assess cardiac related hospitalization and death over a 12 month period by examining medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to perform a 6-minute walk task, with or without use of a cane or walker (must use the same walking assistance device during each session), and walk under 500 meters during task.
2. Symptoms of chronic heart failure for at least 3 months.
3. Clinically stable- defined as not having been hospitalized for a 3 month period, on stable doses of neurohormonal blocking agents and diuretics for at least 3 months.
4. ACC/AHA stages B and C
5. Ability to perform light to moderate exercise (NYHA functional class II and III)
6. Presence of HF with an ejection fraction less than 40%, or diastolic dysfunction
7. Ability to give informed consent
8. At least18 years of age

Exclusion Criteria:

1. History of recent myocardial infarction (1 month)
2. Angina not adequately managed with nitrates.
3. Aortic or mitral stenosis
4. Coronary revascularization, mitral valve repair or any other cardiac surgery or implantation of a biventricular pacemaker within the past 6 months.
5. Severe COPD
6. Recent stroke or significant cerebral neurologic impairment.
7. Active Suicidality
8. Currently participating in an exercise program.
9. Currently taking mood stabilizers (e.g. lithium), benzodiazepines or antipsychotics.
10. Medications (steroids) and medical conditions affecting immune status not limited to Grave's Disease, Rheumatoid Arthritis, Hashimoto's Disease, Sjogren's Disease, Lupus, Multiple Sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (%LVEF) | Change from Baseline in %LVEF Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in cardiac functional capacity as measured by %LVEF on echocardiogram.
End Systolic Volume (ESV) | Change from Baseline in ESV Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in cardiac functional capacity as measured by ESV on echocardiogram.
End Diastolic Volume (EDV) | Change from Baseline in EDV Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in cardiac functional capacity as measured by EDV on echocardiogram.

SECONDARY OUTCOMES:
B-type Natriuretic Peptide (BNP) | Change from Baseline in BNP Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in cardiac functional capacity as measured by serum levels of BNP.
Six-Minute Walk Task (6MWT) | Change from Baseline in 6MWT Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in cardiac functional capacity as measured by 6MWT at post-treatment.
Work Performed on Bicycle Ergometer Task (Watts) | Change from Baseline in Watts Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in cardiac functional capacity as measured by average watts on a mild, graded exercise task on a bicycle ergometer at post-treatment assessment.
Average Number of Steps Across 3 Days (Steps) | Change from Baseline in Steps Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in cardiac functional capacity as measured by the average number of steps measured using a pedometer over a 3 day period immediately following 16 weeks of treatment.
Beck Depression Inventory (BDI) at Post-Treatment | Change from Baseline in BDI Scores Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in depression scores as measured by the BDI immediately following 16 weeks of treatment.
BDI at 8-Week Follow-Up | Change from Baseline in BDI scores at 8-week follow-up
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in depression scores as measured by the BDI at the 8-week follow-up assessment.
BDI at 1-Year Follow-Up | Change from Baseline in BDI Scores at 1-year follow-up
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in depression scores as measured by the BDI at the 1-year follow-up assessment.
Pittsburgh Sleep Quality Inventory (PSQI) at Post-Treatment | Change from Baseline on the (PSQI) Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in sleep quality scores as measured by the PSQI immediately following 16 weeks of treatment.
PSQI at 8-Week Follow-Up | Change from Baseline in PSQI scores at 8-week follow-up
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in sleep quality scores as measured by the PSQI at the 8-week follow-up assessment.
PSQI at 1-Year Follow-Up | Change from Baseline in PSQI Scores at 1-year Follow-Up Assessment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in sleep quality scores as measured by the PSQI at the 1-year follow-up assessment.
Multidimensional Fatigue Symptom Inventory (MFSI) at Post-Treatment | Change from Baseline in MFSI Scores Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in fatigue scores as measured by the MFSI immediately following 16 weeks of treatment.
MFSI at 8-Week Follow-Up | Change From Baseline in MFSI Scores at 8-week Follow-up Assessment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in fatigue scores as measured by the MFSI at the 8-week follow-up assessment.
MFSI at 1-Year Follow-Up | Change From Baseline in MFSI Scores at the 1-Year Follow-Up Assessment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in fatigue scores as measured by the MFSI at the 1-year follow-up assessment.
Minnesota Living with Heart Failure Questionnaire (MLHFQ) at Post-Treatment | Change from Baseline in MLHFQ Scores Immediately Following 16 Weeks of Treatment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in health-related quality of life scores as measured by the MHLFQ immediately following 16 weeks of treatment.
MHLFQ at 8-Week Follow-Up | Change from Baseline in MHLFQ at 8-Week Follow-Up Assessment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in health-related quality of life scores scores as measured by the PSQI at the 8-week follow-up assessment.
MHLFQ at 1-Year Follow-Up Assessment | Change from Baseline in MHLFQ Scores at 1-year Follow-Up Assessment
  Determine whether Tai Chi compared with Resistance Exercise and Health Education control condition will lead to a greater improvement in health-related quality of life scores as measured by the MHLFQ at the 1-year follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura S Redwine, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of Califoria, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Redwine LS, Pung MA, Wilson K, Bangen KJ, Delano-Wood L, Hurwitz B. An exploratory randomized sub-study of light-to-moderate intensity exercise on cognitive function, depression symptoms and inflammation in older adults with heart failure. J Psychosom Res. 2020 Jan;128:109883. doi: 10.1016/j.jpsychores.2019.109883. Epub 2019 Nov 26. PMID 31786338